CLINICAL TRIAL: NCT02082197
Title: A Multicenter, Open-Label, Efficacy and Safety Study of ABT-SLV176 for the Treatment of Hypogonadal Men
Brief Title: An Efficacy and Safety Study of ABT-SLV176 for the Treatment of Hypogonadal Men
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Other - not a safety issue
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-886
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Hypogonadism; Testosterone Deficiency
Keywords: low testosterone
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-SLV176 (Experimental): ABT-SLV176 administered daily
  Interventions: Drug: ABT-SLV176

INTERVENTIONS:
Drug: ABT-SLV176 — ABT-SLV176 administered daily

SUMMARY:
This is an open-study with a 26 week open label treatment period followed by an optional 26 week open label extension. The total treatment period will be 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

Low testosterone

Exclusion Criteria:

* Normal testosterone levels
* Elevated Prostatic Specific Antigen (PSA)
* History of breast or prostate cancer

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with serum total testosterone average concentration, Cavg(0-24) | At Week 12
  Cavg (0-24) is the time-averaged Concentration Over the Dosing Interval of 24 Hours.

SECONDARY OUTCOMES:
Percentage of subjects falling within the pre-defined ranges of maximum total testosterone concentration (Cmax) | At Week 2, Week 4, Week 12 and Week 52
  Cmax is the maximum concentration.
Average serum total testosterone and Dihydrotestosterone (DHT) concentration (Cavg) | At Week 2, Week 4, Week 12 and Week 52
  Cavg is the average concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miller, PharmD, Study Director — AbbVie
Locations (42):
- United States (42):
  - Site Reference ID/Investigator# 124163, Birmingham, Alabama
  - Site Reference ID/Investigator# 123938, Huntsville, Alabama
  - Site Reference ID/Investigator# 125782, Mesa, Arizona
  - Site Reference ID/Investigator# 124157, Phoenix, Arizona
  - Site Reference ID/Investigator# 123937, Tucson, Arizona
  - Site Reference ID/Investigator# 123948, Anaheim, California
  - Site Reference ID/Investigator# 124164, Los Angeles, California
  - Site Reference ID/Investigator# 123920, Los Gatos, California
  - Site Reference ID/Investigator# 124038, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 126202, Denver, Colorado
  - Site Reference ID/Investigator# 123927, Middlebury, Connecticut
  - Site Reference ID/Investigator# 123947, Clearwater, Florida
  - Site Reference ID/Investigator# 123929, Jacksonville, Florida
  - Site Reference ID/Investigator# 123940, Ocala, Florida
  - Site Reference ID/Investigator# 124166, Orlando, Florida
  - Site Reference ID/Investigator# 123945, Ponte Vedra Beach, Florida
  - Site Reference ID/Investigator# 123930, Dunwoody, Georgia
  - Site Reference ID/Investigator# 124395, Wichita, Kansas
  - Site Reference ID/Investigator# 125784, Crestview Hills, Kentucky
  - Site Reference ID/Investigator# 123919, Lexington, Kentucky
  - Site Reference ID/Investigator# 123925, Baltimore, Maryland
  - Site Reference ID/Investigator# 123936, Methuen, Massachusetts
  - Site Reference ID/Investigator# 124160, Las Vegas, Nevada
  - Site Reference ID/Investigator# 123939, Las Vegas, Nevada
  - Site Reference ID/Investigator# 123932, Lawrenceville, New Jersey
  - Site Reference ID/Investigator# 123943, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 123926, Garden City, New York
  - Site Reference ID/Investigator# 125783, New York, New York
  - Site Reference ID/Investigator# 123928, Poughkeepsie, New York
  - Site Reference ID/Investigator# 124165, Charlotte, North Carolina
  - Site Reference ID/Investigator# 123933, Morehead City, North Carolina
  - Site Reference ID/Investigator# 123921, Salisbury, North Carolina
  - Site Reference ID/Investigator# 124162, Cleveland, Ohio
  - Site Reference ID/Investigator# 123917, Bala-Cynwyd, Pennsylvania
  - Site Reference ID/Investigator# 123931, Jenkintown, Pennsylvania
  - Site Reference ID/Investigator# 123924, Greer, South Carolina
  - Site Reference ID/Investigator# 123895, Chattanooga, Tennessee
  - Site Reference ID/Investigator# 123946, Nashville, Tennessee
  - Site Reference ID/Investigator# 123923, Austin, Texas
  - Site Reference ID/Investigator# 123922, Dallas, Texas
  - Site Reference ID/Investigator# 124167, Dallas, Texas
  - Site Reference ID/Investigator# 123944, San Antonio, Texas